CLINICAL TRIAL: NCT04099524
Title: Effectiveness of a Non-Invasive, Low-Intensity Brain Stimulation Approach in Addressing Emotional Regulation
Brief Title: CogT BEEM Study (a tDCS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Vankee Lin, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00003664; R21MH120734 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Neuropsychiatric Syndrome
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Experimental): We will apply the stimulation for 20 minutes using current at 1.5mA with a ramp up and ramp down period of 30 seconds at the start and end of the session.
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): tDCS will ramp up for 30 seconds with 1 mA current and then ramp off within 10 seconds. As 30 seconds is too short for tDCS to have any effects, this will be the control condition. tDCS is on for 30 seconds because that is usually the only time individuals would experience tingling and itching - a factor we aim to equate between experimental and control conditions.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS (LPG/C3-anode, orbitofrontal cortex/Fp2-cathode) will be administered for 4 weeks (1 session per weekday for 2 weeks, and then 2 sessions per week for 2 weeks, for a total of 14 sessions). All subjects will receive anodal tDCS stimulation for 20 minutes per session, on C3 and the cathode electrode on Fp2 using 10/20 EEG system. tDCS will be applied with a pair of 35 cm2 single-use sponges soaked in approximately 4mL of saline solution on each side (~8mL per sponge) connected to the stimulator. During the 20-minute tDCS session, we will use online tDCS design (i.e., a subject will simultaneously work on the visual attention-oriented task.

SUMMARY:
Co-existing neuropsychiatric symptoms (NPS) in patients with mild cognitive impairment (MCI), especially those worsening over time, are associated with more rapid cognitive and functional decline and a greater risk of Alzheimer's disease (AD). Optimal NPS management, meaning effectively managing multiple NPS simultaneously, requires a solid understanding of the shared neural mechanism across NPS. The goal of this proof-of-concept mechanistic intervention study is to validate the causal relationship between a NPS-shared neural circuit the investigators previously discovered and various NPS. The investigators will modify a key region within the NPS-shared neural circuit [i.e. left precentral gyrus (LPG), critical for regulating visual attention] with anodal transcranial direct current stimulation (tDCS). Our central hypothesis is that an activation of LPG and a reorganization of NPS-shared neural circuit will link to improvement in multiple NPS. Using a Stage 0 pilot randomized control trial design the investigators will recruit n = 40 older adults with informant-rated NPS that has worsened in the past 2 years, which is considered the most detrimental type of NPS in MCI. The investigators will assign participants to 4-week active anodal vs. sham LPG online tDCS group. The investigators will assess resting-state and visual attention task-related functional MRI and informant-rated NPS at baseline, and the end of week 4 and week 8, and diffusion MRI at baseline. The two primary aims are to determine the effect of tDCS on NPS-shared neural circuit (Aim 1), as well as the relationship between NPS-shared neural circuit and informant-report NPS (Aim 2). The exploratory aim will be to examine the relationship between NPS and the coherence between structural and functional aspects of the NPS-shared neural circuit. Probing the LPG via anodal tDCS provides a way to experimentally test the causal relationship between our previously discovered NPS-shared neural circuit and informant-rated NPS. The proposed research is highly innovative, while scientifically grounded, for targeting one brain region that may affect multiple NPS. Validating the hypotheses has the potential for future R01 study that directly conducts a Stage 2 trial addressing NPS in MCI, and thus ultimately improves patient's quality of life and reducing caregiving burden.

ELIGIBILITY:
Inclusion Criteria:

1. Forty subjects with MCI and comorbid NPS, which have worsened in the past 2 years (as rated by their study-partner's responses to the NPI-Q):

1. In the past month, presence of > 2 symptoms; and
2. Compared to two years ago, having > 1 pre-exist symptom whose severity rating has worsened, or having > 1 new symptom; 2. Consensus diagnosis of "mild cognitive impairment due to Alzheimer's disease" based on 2011 NIA-AA diagnostic criteria by the investigators based on screening information: i. Memory deficits at screening: 1 standard deviation (SD) below age- and/or education- corrected population norms for the Rey Auditory Verbal Learning Test (RAVLT, Lists C&D); ii. Global memory deficits at screening: Montreal Cognitive Assessment (MoCA, Version 2) total score within the range 18 ≤ x ≤ 26, after educational adjustment; iii. Preserved activity of daily living: ADL-PI-self total score ≤ 30; iv. Absence of dementia. 3. Stable (same dosage, frequency, type) on memory medications for ≥ 3 months before screening; 4. Stable (same dosage, frequency, type) on any anti-depressants, antipsychotics, and/or anxiolytics for ≥ 7 days; 5. Community-dwelling: Subjects live in homes or independent- and assisted- living facilities (i.e. - not nursing home residents, due to the large cognitive variability in nursing home residents); 6. Aged 60-89 years at screening; 7. English-speaking; 8. Adequate visual and hearing acuity for testing; 9. Verified tDCS and MRI safety: Subject should not have any contraindications to either and pass safety screening questions for both (see exclusion section for more information); 10. Capacity to consent, based on responses and ratings to the UCSD Brief Assessment of Capacity to Consent (UBACC) form modified for this study 11. Availability of a study partner who spends at least several hours per week with the subject, supervises his/her care, and who is willing to accompany the subject to some study visits and participate in the study; 12. Informed consent for study participation obtained by both the subject and his/her study partner; 13. Agree to donate 20mL of blood at baseline, after fasting for at least 8 hours (only water and prescribed medicines)

Exclusion Criteria:

* Participants may be excluded from enrollment, or have their enrollment deferred until they are eligible, for the reasons listed below. Final decisions regarding enrollment will be determined by the PI on a case-by-case basis.

  1. Presence of any neurological or vascular disorders (e.g. - Multiple Sclerosis [MS], Traumatic Brain Injury [TBI], chronic heart failure [CHF], Parkinson's disease [PD]);
  2. Clinical diagnosis of dementia as defined by the most recent version of the DSM;
  3. Current enrollment in another study aimed at improving cognitive abilities and/or emotional well-being;
  4. MRI contraindications (e.g. - pacemaker, implantable cardioverter defibrillator [ICD], aneurysm clips, severe claustrophobia);
  5. tDCS contraindications (e.g. - scalp or skin condition, history of migraines, seizures or epilepsy, and/or strokes, TBI), metallic implants, history of adverse effects to previous tDCS or other brain stimulation techniques).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cabin, Ur, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turnbull A, Anthony M, Tadin D, Porsteinsson AP, Heffner K, Lin FV. Effect of online tDCS to left somatomotor cortex on neuropsychiatric symptoms among older adults at risk for dementia. Cortex. 2023 Feb;159:131-141. doi: 10.1016/j.cortex.2022.10.015. Epub 2022 Dec 17. PMID 36623419

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: all participants enrolled were assigned to groups.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: We conducted group comparisons of baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6.6) | 73 (7.1) | 71 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White, Non-Hispanic/Latino | 19 | 19 | 38
  Race: White, Hispanic/Latino | 0 | 1 | 1
  Race: African American/Black | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change of C3 Activation (NPS-shared Neural Circuit Measure
Description: Change of arbitrary unit LPG activation in response to visual attention task (measured using task related fMRI). No theoretical minimum or maximum exists for this scale.
Time Frame: from baseline to post-intervention (4 weeks)
Population: AR(1) covariance matrix with Generalized Estimating Equation (GEE) model. Data from 35 subjects (18 from intervention and 17 from control) were included in the data analysis on LSMC: in addition to the one participant that withdrew, one participant's data was excluded for excessive motion during MRI scanning, two for issues with co-registration and normalization, and one did not complete MRI scanning at timepoint 2 due to claustrophobia.
Measure: Mean (Standard Deviation); unit: change of arbitrary unit LPG activation
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 17
change of arbitrary unit LPG activation | -0.15 (0.39) | 0.01 (0.33)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Test type: Superiority — The analysis was based on evaluating whether active tDCS is superior than sham tDCS on outcomes; p < 0.05, Mixed Models Analysis — multiple correction adjusted p<0.05; Mean Difference (Final Values) = -0.18
Statistical Analysis 2: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p < 0.05, Mixed Models Analysis — multiple correction adjusted p<0.05; Mean Difference (Final Values) = 0.20

2. Secondary Outcome: Change of Patient-report NPS
Description: Patient-reported NPS was measured using three mood-related questionnaires that probed mood within the past week: depression (Geriatric Depressive Scale ;GDS-30); anxiety (State-Trait-Anxiety-Inventory; STAI-state); and apathy (Apathy Evaluation Scale; AES). Total scores from individual measures were z-transformed (higher score indicating severer symptoms) across timepoints and averaged to create a composite mood score. A Z-score of 0 represents the population mean. Change of Z-score from baseline to post-intervention was used.
Time Frame: from baseline to post-intervention (4 weeks)
Population: AR(1) covariance matrix with Generalized Estimating Equation (GEE) model; 1 person from control gorp was withdrawn during the beginning of intervention.
Measure: Mean (Standard Deviation); unit: change of Z-score
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 19
change of Z-score | -0.22 (0.52) | -1.01 (2.52)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Test type: Superiority — The analysis was based on evaluating whether active tDCS is superior than sham tDCS on outcomes; p < 0.05, Chi-squared; chi-square = 3.14

3. Primary Outcome: Change of C3 Connectivity (NPS-shared Neural Circuit Measure 21)
Description: Change of arbitrary unit of correlation between LPG and amygdala at rest (resting fMRI). No theoretical minimum or maximum exists for this scale.
Time Frame: from baseline to post-intervention (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change of arbitrary unit LPG correlation
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 17
change of arbitrary unit LPG correlation | 0.10 (0.26) | -0.10 (0.29)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Test type: Superiority — The analysis was based on evaluating whether active tDCS is superior than sham tDCS on outcomes; p < 0.05, Mixed Models Analysis — multiple correction adjusted p<0.05; Mean Difference (Final Values) = 0.20

4. Secondary Outcome: Change of Informant-rated NPS
Description: Informant-reported NPS was measured using the 12-domain Neuropsychiatric Inventory (NPI-Full), including both frequency and severity (based on present symptoms) during the past week. We first calculated the frequency x severity for each domain, then averaged across domains, and finally adjusted for caregiving burden. Higher is worse. We calculated the change of the arbitrary score from baseline to post-intervention. No theoretical minimum and maximum scores exist
Time Frame: from baseline to post-intervention (4 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change of arbitrary score
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 19
change of arbitrary score | -0.04 (0.45) | -0.87 (1.63)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; Test type: Superiority — The analysis was based on evaluating whether active tDCS is superior than sham tDCS on outcomes; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.84

ADVERSE EVENTS:
Time Frame: 25 months
Description: The definitions of adverse events or serious adverse events are the same as defined in the clinicaltrial.gov definitions.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT04099524/Prot_SAP_000.pdf